CLINICAL TRIAL: NCT06237959
Title: A 24-Week, Randomized, Double-blind, Placebo-controlled Clinical Study to Evaluate the Efficacy and Safety of Proso Millet and Wheat Extract(Keranat™) on Hair Health
Brief Title: Evaluate the Efficacy and Safety of Proso Millet and Wheat Extract(Keranat™) on Hair Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nutracore (Industry)
Collaborators: Novarex (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NC07-NOVA-2022
Record Dates: First submitted 2024-01-02; First posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Hair Damage
Keywords: Hair gloss; Hair elasticity; Hair strength; Hair thickness; Anagen hair; Number of hair loss

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Keranat™ (Experimental): Keranat™ capsule will be administered orally twice daily for 24 weeks.
  Interventions: Dietary Supplement: Keranat™
- Placebo (Placebo Comparator): Placebo capsule will be administered orally twice daily for 24 weeks.
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Keranat™ — 300 mg/capsule(proso millet and wheat extract 600 mg/day)
  Arms: Keranat™
Dietary Supplement: placebo — 300 mg/capsule(600 mg/day as placebo)
  Arms: Placebo

SUMMARY:
The purpose of this randomized, double-blind, placebo-controlled study will be to evaluate whether the daily intake of Keranat™ for 24 weeks can promote the gloss and elasticity of hairs, improve their density and strength, and reduce hair loss.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 and 60
* Hair gloss score of 3 or less and a hair damage score of less than 18 according to the visual evaluation classification method.
* Willing to maintain the same hairstyle, hair color, hair length, and hair regimen throughout the study period.
* Subject must be able to comprehend and voluntarily sign study procedures and consent forms.

Exclusion Criteria:

* Those diagnosed with and receiving treatment for the alopecia within 3 months before screening(androgenetic alopecia, alopecia areata, Telogen effluvium, etc.)
* Use of that may affect hair or hair loss symptoms treatment medicine, dietary supplements, or treatments containing herbal medicine ingredients within 3 months before screening.
* Any active scalp or skin disease that may interfere with the study treatment and evaluations.
* Pregnancy or breastfeeding or planning pregnancy
* Case of abnormal values at creatinine (excess at the upper limit of the reference range)
* Case of abnormal values at ALT or AST (2 times excess at the upper limit of the reference range)

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2022-11-02 (Actual); Primary Completion 2023-06-12 (Actual); Study Completion 2023-12-11 (Actual)

PRIMARY OUTCOMES:
The change of hair elasticity | Change of the week 24 from baseline
  To evaluate the change in hair elasticity between the Keranat™ and placebo group.
  Hair elasticity was measured using an Expert 7601Tension Testing System.
The change of hair gloss | Change of the week 24 from baseline
  To evaluate the change in hair gloss between the Keranat™ and placebo group. Hair gloss was measured using a Skin-Glossy meter GL200.

SECONDARY OUTCOMES:
The change of hair thickness | Change of the week 24 from baseline
  To evaluate the change in hair thickness improvement between the Keranat™ and placebo group. Hair thinness was assessed by measuring hair diameter using a microscope and ToupLite software.
The change of anagen hair ratio(%) | Change of the week 24 from baseline
  To evaluate the change in the ratio of anagen hair between the Keranat™ and placebo group. Changes in Hair growth that occurred in the hair removal area for 3 days were analyzed using the Image-Pro® 10 program.
The change in hair loss amount | Change of the week 24 from baseline
  To evaluate the change in the number of hair loss between the Keranat™ and placebo group. Collected and counted the number of lost hair.
The change of number of hair per unit area | Change of the week 24 from baseline
  To evaluate the change in the number of hairs per unit area between the Keranat™ and placebo group. The number of hairs per unit area of the hair removal area was counted using Folliscope PS.
The change of hair distribution score through clinical photography | Change of the week 24 from baseline
  To evaluate the change in hair distribution score through clinical photography between the Keranat™ and placebo group before and after intake. This evaluates improvement and deterioration on a 7-point scale, with higher scores meaning improvement. By comparing photos before and after intake, if there is no change, 0 points, improvement is a maximum of 3 points, and worsening is a minimum of -3 points.
Self-reported Hair health assessments | Change of the week 24 from baseline
  To evaluate the change in Hair health improvement between the Keranat™ and placebo group. The evaluation was conducted through Patient Report Outcome(PRO) using a standardized survey form. Survey allowing for participant-report changes in hair health as a result of intervention using a 7-point scale.
The change of serum levels of cytokines (IL-1, TNF-α, PGE2) | Change of the week 24 from baseline
  To evaluate the change in serum levels of cytokines through clinical photography between the Keranat™ and placebo group.

CONTACTS AND LOCATIONS:
Locations (1):
- KSRC Korean Skin Research Center, Seongnam-si, Gyeonggido, South Korea

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-01): https://cdn.clinicaltrials.gov/large-docs/59/NCT06237959/Prot_SAP_000.pdf